CLINICAL TRIAL: NCT02786719
Title: A Safety Pilot Study of High Risk Induction Chemotherapy for Neuroblastoma Without Prophylactic Administration of Myeloid Growth Factors
Brief Title: High-Risk Neuroblastoma Chemotherapy Without G-CSF
Acronym: SPRING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Sarah Whittle, Instructor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-38179 (SPRING); SPRING (Other: Baylor College of Medicine)
Record Dates: First submitted 2016-05-23; First posted 2016-06-01 (Estimated); Results first posted 2020-03-12 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Neuroblastoma
Keywords: Sargramostim; Cyclophosphamide; Topotecan; Cisplatin; Dexrazoxane; Doxorubicin; Etoposide; Filgrastim; Vincristine; Mesna
MeSH Terms: conditions — Neuroblastoma | interventions — Topotecan; Cyclophosphamide; Cisplatin; Etoposide; Vincristine; Doxorubicin; sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Neuroblastoma treatment without G-CSF (Experimental): Induction chemotherapy only, including 6 cycles of chemotherapy, tumor resection, and stem cell collection
  Interventions: Drug: Topotecan; Drug: Cyclophosphamide; Drug: Cisplatin; Drug: Etoposide; Drug: Vincristine; Drug: Doxorubicin; Drug: Sargramostim

INTERVENTIONS:
Drug: Topotecan — CYCLE 1+2 (given by intravenous catheter daily for 5 days)
  Other Names: hycamtin
Drug: Cyclophosphamide — CYCLE 1+2 (given by intravenous catheter daily for 5 days)
  Other Names: Cytoxan
Drug: Cisplatin — Cycle 3+5 (given daily x 4 days)
  Other Names: CDDP; Platinol
Drug: Etoposide — Cycle 3+5 (given daily for 3 days)
Drug: Vincristine — Cycle 4+6 (given daily for 3 days)
  Other Names: Oncovin
Drug: Cyclophosphamide — Cycle 4+6 (given daily for 2 days)
  Other Names: Cytoxan
Drug: Doxorubicin — Cycle 4+6 (given daily for 3 days)
  Other Names: Adriamycin
Drug: Sargramostim — Granulocyte macrophage colony stimulating factor (rhu GM-CSF, rGM-CSF, GM-CSF)
  Other Names: GM-CSF

SUMMARY:
Patients will be asked to participate in this study because patients have been diagnosed with high-risk neuroblastoma, a common childhood cancer which has aggressive features. If left untreated, high-risk neuroblastoma is fatal. Children with high-risk neuroblastoma often respond to current available treatments, but there is a high risk that the cancer will return.

This study will test the safety of giving standard induction treatment for high-risk neuroblastoma without one of the drugs commonly used to prevent side effects. Current treatment for high-risk neuroblastoma includes anti-cancer drugs (chemotherapy), surgery, radiation therapy and high-dose chemotherapy with hematopoietic stem cell rescue. Treatment takes about one year to complete and occurs in 3 phases: induction, consolidation, and maintenance. This study is limited to the induction phase of treatment.

Induction therapy includes six chemotherapy drugs given in different combinations every 3 weeks for a total of 6 courses. For the past decade, induction chemotherapy has been followed by a drug called granulocyte colony stimulating factor (G-CSF, filgrastim, peg-filgrastim, Neupogen, or Neulasta) to prevent side effects from the chemotherapy. G-CSF is routinely given to patients with high risk neuroblastoma after chemotherapy to stimulate white blood cell production and shorten the time period when the absolute neutrophil count (ANC), a type of white blood cell, is low after chemotherapy. G-CSF is known to shorten the period of low ANC by approximately 3 days. When the ANC is lowest, a patient is most at risk of getting a bacterial infection.

Recent lab experiments in mice have shown that neuroblastoma tumor cells may respond to G-CSF by growing faster and metastasizing (spreading to other parts of the body). There have been no clinical trials comparing the survival of children with high risk neuroblastoma with or without G-CSF. This clinical trial is the first step towards giving induction chemotherapy with less G-CSF.

The goal of this study is to determine if it is safe to give induction chemotherapy to children with neuroblastoma without giving G-CSF routinely.

DETAILED DESCRIPTION:
Chemotherapy:

CYCLE 1+2: Topotecan and cyclophosphamide

Cycle 3+5: Cisplatin and Etoposide

Cycle 4+6: Vincristine, Cyclophosphamide and Doxorubicin

Stem cell collection: After the third cycle of chemotherapy, stem cells will be collected for possible stem cell transplantation at a later date using apheresis. In order to have enough stem cells present in the blood, the patient will need to receive daily G-CSF injections before this collection.

Surgery: After the 5th cycle of chemotherapy, most patients will have surgery to remove as much remaining tumor as possible.

Growth factor support: Growth factors to increase the number of white blood cells, G-CSF and GM-CSF(granulocyte-macrophage colony stimulating factor) will not be given routinely in this study. GM-CSF will be given for patients who have serious bacterial infections or delays in administering chemotherapy because of low neutrophil counts. All people enrolled on the study will receive GM-CSF prior to having surgical removal of the main tumor. All people enrolled on the study will also receive G-CSF prior to having patients stem cells collected.

Optional survey: This research study includes an optional survey regarding quality of life while on the study. This survey will be filled out after cycles 1 and 4 of chemotherapy.

Drug Shortages:

In the event of a drug shortage of a medication that is not a G-CSF or GM-CSF product, the provider may use best clinical judgment regarding omission of the agent or substitution with a different agent. The medical and research records of study patients should reflect that the patient was informed of any delays and/or modifications in protocol therapy related to the shortage of the agent and the associated risks.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 12 months and less than 18 years old at diagnosis
* Newly diagnosed neuroblastoma or ganglioneuroblastoma as verified by histology and/or demonstration of tumor cells in bone marrow with elevated urinary catecholamine metabolites
* Must meet criteria for High Risk disease

  * Patients with International Neuroblastoma Staging System (INSS) stage 4 disease are eligible with the following: MYCN gene amplification (greater than four-fold increase in MYCN signals as compared to reference signals), regardless of age or additional biologic features, Age greater than 18 months ( greater than 547 days) regardless of biologic features, Age 12 -18 months (365 - 547 days) with any of the following unfavorable biologic features (unfavorable pathology and/or DNA index = 1) or any biologic feature that is indeterminate/unsatisfactory/unknown
  * Patients with INSS stage 3 disease are eligible with the following: MYCN amplification, regardless of age or additional biologic features, Age greater than 18 months ( greater than 547 days) with unfavorable pathology, regardless of MYCN status
  * Patients with INSS stage 2a/2b with MYCN amplification regardless of age or additional biologic features
  * Patients greater than or equal to 365 days initially diagnosed with INSS stage 1 or 2 who progressed to a stage 4 without interval chemotherapy
* Patients may have had no prior systemic therapy except: Localized emergency radiation to sites of life threatening or functioning disease, No more than 1 cycle of chemotherapy according to low or intermediate risk regimens prior to determination of MYCN amplification and histology, as long as the patient DID NOT receive any type of granulocyte colony stimulating factor (G-CSF) as part of that therapy.
* Patients must have adequate hematopoietic function defined as: Absolute neutrophil count (ANC) greater than or equal to 750/μL, Platelet count greater than or equal to 75,000/μL, The above criteria do not have to be met if the patient has bone marrow involvement of tumor.
* Patients must have adequate liver function defined as: Direct bilirubin less than or equal to 1.5 mg/dL or total bilirubin ≤ 1.5 mg/dL, aspartate aminotrasnferase (AST) and alanine aminotransferase (ALT) less than or equal to10 x upper limit of normal for age
* Patients must have adequate renal function as defined as: Creatinine clearance (CrCl) or radioisotope glomerular filtration rate (GFR) greater than or equal to 70 mL/min/.73 m2 OR A serum creatinine based on age/gender.
* Patients must have adequate cardiac function as defined as: Shortening fraction of greater than or equal to 27 % by echocardiogram, or Ejection fraction of greater than or equal to 50 % by radionuclide angiogram

Exclusion Criteria:

* Patients who do not meet inclusion criteria
* Patients who are pregnant or lactating
* Patients who have received G-CSF since the time of diagnosis of the current disease

Ages: 12 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2016-06; Primary Completion 2019-02-05 (Actual); Study Completion 2019-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Whittle, MD, BA, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Rady Children's Hospital, San Diego, California
  - Texas Children's Hospital, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- High Risk Neuroblastoma Patients: This was a single arm study- all participants enrolled in single arm which provided 6 cycles of chemotherapy without prophylactic G-CSF for 4 cycles (1,2,4 and 6), and with G-CSF for stem cell collection after cycle 3, and GM-CSF administration after cycle 5 in preparation for surgical resection.
Period: Overall Study
Arm/Group | High Risk Neuroblastoma Patients
Started | 13
Completed | 12
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: all participants evaluable for infection endpoint
Groups:
- Single Arm: Single arm study- all participants enrolled in single arm
Arm/Group | Single Arm
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 2.9 [1.1 to 6.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 7
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 12
International Neuroblastoma Risk Group Stage [Count of Participants; unit: Participants]
  L2 (localized with image defined risk factors) | 2
  M (metastatic) | 10
MYCN gene amplification [Count of Participants; unit: Participants] — Amplification of MYCN gene, a poor prognostic factor in neuroblastoma
  Participants
    Yes | 6
    No | 6
Marrow involvement [Count of Participants; unit: Participants]
  Yes | 9
  No | 3

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Infection
Description: Incidence of infections in chemotherapy cycles NOT followed by hematopoietic growth factors
Time Frame: through study completion, approximately 5 months
Population: Includes all patients evaluable for endpoint
Measure: Number; unit: infections
Groups:
- High Risk Neuroblastoma Patients: Single arm study- all participants enrolled in single arm
Arm/Group | High Risk Neuroblastoma Patients
Number analyzed (Participants) | 12
infections | 6

2. Secondary Outcome: Delay in Chemotherapy Administration Due to Prolonged Neutrophil Recovery
Description: incidence of delay in chemotherapy administration due to prolonged neutrophil recovery
Time Frame: through study completion, approximately 5 months
Population: 58 cycles of chemotherapy administered to 12 participants
Measure: Number; unit: chemotherapy cycles
Units Other Than Participants: Chemotherapy cycles
Arm/Group | High Risk Neuroblastoma Patients
Number analyzed (Participants) | 12
Number analyzed (Chemotherapy cycles) | 58
chemotherapy cycles | 9

3. Secondary Outcome: the Response Rate Following Induction Chemotherapy Without Prophylactic Granulocyte Colony Stimulating Factor (G-CSF)
Description: Response rate in the participants that completed all 6 cycles of induction chemotherapy on study. Response rate as categorize by International neuroblastoma response criteria.
  * Complete response (CR): No evidence of primary tumor; no evidence of metastases (chest, abdomen, liver, bone, bone marrow, nodes, etc.), and urine catecholamines homovanillic acid (HVA)/ vanillylmandelic acid (VMA) normal. MIBG scan must be negative to qualify for CR.
  * Very good partial response (VGPR): Greater than 90% reduction in primary tumor; no metastatic tumor (as above except bone); no new bone lesions, all pre-existing lesions improved, HVA/VMA normal
  * Partial Response (PR): 50-90% reduction of primary tumor; 50% or greater reduction in measurable sites of metastases; 0-1 bone marrow samples with tumor; number of positive bone sites decreased by 50%
Time Frame: through study completion, approximately 5 months
Population: Completed all 6 cycles of induction chemotherapy on study
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Neuroblastoma Patients
Number analyzed (Participants) | 8
Participants
  Partial response | 2
  Very good partial response | 2
  Complete Response | 4

ADVERSE EVENTS:
Time Frame: Reporting period for each patient was from enrolling on trial until ANC recovery >750 from final cycle of chemotherapy administered while patient on study (max of 6 cycles).
Description: A systematic assessment was performed using regular laboratory assessment as well as regular investigator assessment of clinical records for AEs.
  All-Cause Mortality was assessed for all 13 participants who signed the informed consent. Serious and Other (Not Including Serious) Adverse Events were only assessed for the 12 participants who received treatment.
Arm/Group | High Risk Neuroblastoma Patients
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 11/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High Risk Neuroblastoma Patients (N=12)
Febrile Neutropenia (Blood and lymphatic system disorders) | 9
bacteremia (Infections and infestations) | 4
Skin/soft tissue infection (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Sinusoidal obstruction syndrome (Hepatobiliary disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Risk Neuroblastoma Patients (N=12)
ALT increased (Hepatobiliary disorders) | 1 (1) — Alanine aminotransferase increased
Alk phos increased (Hepatobiliary disorders) | 1 (1) — Alkaline phosphatase increased
Anemia (Blood and lymphatic system disorders) | 12 (73) — Anemia
AST increased (Hepatobiliary disorders) | 1 (1) — Aspartate aminotransferase increased
Neutropenia (Blood and lymphatic system disorders) | 12 (100) — Neutrophil count decreased
Pain (Musculoskeletal and connective tissue disorders) | 2 (2) — Pain in extremity
Thrombocytopenia (Blood and lymphatic system disorders) | 12 (93) — Platelet count decreased
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Pleural effusion
Rash (Skin and subcutaneous tissue disorders) | 1 (1) — Rash
Weight loss (General disorders) | 1 (1) — Weight loss
WBC decreased (Blood and lymphatic system disorders) | 12 (119) — White blood cell decreased

LIMITATIONS AND CAVEATS:
This study was designed to pilot safely decreasing exposure to G-CSF. To formally test the non-inferiority of not giving G-CSF a much larger sample size would be needed. This study does not conclude that G-CSF prevents infections.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-14): https://cdn.clinicaltrials.gov/large-docs/19/NCT02786719/Prot_SAP_000.pdf